CLINICAL TRIAL: NCT05658250
Title: Feasibility of CRE8 Polymer-free Amphilimus-eluting sTEnt in Patients With Diffuse Long Lesions (CREATE Trial): Prospective, Observational Study
Brief Title: CREATE Trial, Prospective, Observational Study
Status: Active, not recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Collaborators: Dio (Industry)
Responsible Party: Principal Investigator, Deok-Kyu Cho, Professor, Yonsei University
Other Study IDs: 9-2021-0093
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Drug Eluting Stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CRE8 polymer-free Amphilimus-eluting stent, Cre8 evo stent — Percutaneous coronary intervention using a Cre8 stent, Cre8 evo stent for long lesions

SUMMARY:
Observation of the safety and effectiveness of Cre8 stent, Cre8 evo stent in patients with ischemic heart disease with long coronary lesions

DETAILED DESCRIPTION:
The purpose of this study is to observe the prognosis of 300 patients with long lesions over 30 mm treated with a new-generation Cre8 stent, Cre8 evo stent that is polymer-free and releases fat-soluble ampilimus in the real world. In addition, in the case of inserting a 46mm very long stent through sub-analysis, we also want to check whether stent expansion is performed through OCT rather than IVUS.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years of age or older
2. Clinical evidence of coronary artery disease, including asymptomatic ischemia, stable angina, and acute coronary syndrome (unstable angina, non-ST-segment elevation myocardial infarction, ST-segment elevation myocardial infarction)
3. Coronary artery lesion length 30 mm or more
4. Those who voluntarily agreed in writing to participate in this clinical study

Exclusion Criteria:

1. Remaining life expectancy is less than 1 year
2. Subjects with known hypersensitivity or contraindication to the following drugs or substances: heparin, aspirin, clopidogrel, prasugrel, ticagrelor
3. In case the other researcher judges that it is inappropriate to participate in this study (pregnant women, the elderly, etc.)

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 300 patients underwent Cre 8 stent, Cre8 evo stent implantation of 30 mm or more
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-08-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure including deaht, MI, ST, TLR | 12 months after the index procedure
  number of Target lesion failure including deaht, MI, ST, TLR

SECONDARY OUTCOMES:
All cause death | 12 months after the index procedure
  number of All cause death
Cardiac death | 12 months after the index procedure
  number of Cardiac death
Myocardial infarction | 12 months after the index procedure
  number of Myocardial infarction
Stent thrombosis : definite or probable stent thrombosis by ARC definition | 12 months after the index procedure
  number of Stent thrombosis
Target lesion revascularization | 12 months after the index procedure
  number of Target lesion revascularization
Target vessel revascularization | 12 months after the index procedure
  number of Target vessel revascularization
Stroke | 12 months after the index procedure
  number of Stroke
BARC bleeding 2-5 | 12 months after the index procedure
  number of BARC bleeding 2-5
Stent overexpansion by OCT | immediately after the index procedure in hospitalization
  Maximal stent diameter/ each diameter of stent

CONTACTS AND LOCATIONS:
Locations (1):
- Yongin Severance Hospital, Yongin, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No